CLINICAL TRIAL: NCT01306825
Title: Clinical Evaluation of Daptomycin Bone Penetration
Acronym: DAPTO-HUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4683
Record Dates: First submitted 2011-02-25; First posted 2011-03-02 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-03

CONDITIONS: Bone and Joint Infections
Keywords: Daptomycin; Bone disease,infectious; Osteomyelitis; Diabetic foot; Staphylococcus aureus
MeSH Terms: conditions — Bone Diseases, Infectious; Osteomyelitis; Diabetic Foot; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bone and joint infections are commonly due to Gram-positive bacteria. Treatment of these infections is difficult because of the need of prolonged duration of antimicrobial agents in combination with surgical procedure. Moreover, in recent years, a growing resistance pattern to various antimicrobial agents has been observed for Gram-positive bacteria. Consequently, there is an urgent need for new drugs with high bone penetration for the treatment of those infections. The investigators hypothesized that daptomycin allow to achieve high concentrations in bone compartments.

ELIGIBILITY:
Inclusion criteria:

* Patient under treatment with daptomycin for more than 3 days with dosage at 6 mg/kg
* Patient undergoing imperative surgery with bone withdrawal
* Signed, and dated informed consent as defined by the Institutional Review Board
* Male and female patients older than 18 years of age
* Patients with social insurance
* Patient with information on previous mandatory medical examination

Exclusion criteria :

* Patient with no treatment by daptomycin or with a dosage < 6mg/kg or with less than 3 doses of daptomycine
* Patient with no need for surgery
* Patient younger than 18 years of age
* Pregnant and nursing women
* Patient refusal for inclusion
* Patients with deprived liberty
* Inability to complete the informed consent process because of problems with mental capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient under treatment with daptomycin and undergoing imperative surgery with bone withdrawal
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Patients' percentage of which the intra-osseous daptomycin concentration is ≥ 8 times MIC (if available) or ≥ 8 times critical concentration (if Bacteriological documentation is unavailable) | 5 min before started administration of daptomycin, 5 min after administration of daptomycin and at random after perfusion of daptomycin

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lefebvre, MD, Study Director — Service des maladies infectieuses et tropicales - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg
Locations (3):
- France (3):
  - Service d'Orthopédie - Hôpital Centre de Chirurgie Orthopédie et de la Main (CCOM) - Hôpitaux Universitaires de Strasbourg - 10 av Achille Baumann -, Illkirch-Graffenstaden
  - Plateau Technique de Microbiologie - Hôpitaux Universitaires de Strasbourg - 1, rue Koeberlé, Strasbourg
  - Service des maladies infectieuses et tropicales - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg